CLINICAL TRIAL: NCT01337453
Title: Flu-Like Symptoms as a Complication of Botulinum Toxin Therapy
Status: Completed | Type: Observational
Sponsor: Christine Hunter (Other)
Collaborators: Merz North America, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Christine Hunter, Research Nurse Manager, Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Other Study IDs: H-27678
Record Dates: First submitted 2011-04-14; First posted 2011-04-19 (Estimated); Last update posted 2012-08-24 (Estimated); Status verified 2012-08

CONDITIONS: Flu-like Symptoms
Keywords: botulinum toxin; flu like symptoms; frequency of FLS; Botox

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Flu-like symtoms, incidence: The frequency of FLS will be estimated by number of patients and number of Botox treatments.

SUMMARY:
Botulinum toxin (BoNT) has become a revolutionary treatment for many neurological, autonomic, gastrointestinal, genitourinary, and cosmetic disorders. The use of this treatment requires expertise in dosage calculations and application technique to avoid potential side effects. Most adverse events (AEs) related to BoNT are local and related to its mechanism of action, i.e., paralysis of unwanted muscles. However, systemic AEs may also be observed. Flu-like symptoms (FLS) are well recognized AEs in patients treated with BoNT; however there is a paucity of information regarding the frequency, clinical impact, and associated risk factors of this particular complication.

Between December 1989 and May 2003, 1,437 reports of BoNT-related AEs were registered at the Food and Drug Administration (FDA). FLS were reported in 4.6% of serious, and 3.2% of non-serious side effects.

In this study, the investigators aim to assess prospectively the frequency, clinical characteristics, and risk factors for development of FLS in a group of patients affected with diverse movement disorders and treated with BoNT type A at the Parkinson's Disease Center and Movement Disorders Clinic (PDCMDC) of Baylor College of Medicine (BCM). The investigators will also assess biomarker of inflammatory response in those patients who develop FLS after treatment with BoNT.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with any movement disorder: dystonia, tremor, tics, myoclonus or tardive dyskinesias and treated with botulinum toxin type A (Botox or Dysport) to type B (Myobloc)
2. Patients who will be injected in at least two consecutive visits in our clinic, three months apart.
3. We will invite patients who are regularly treated in our clinic "established patients" and those who will be treated for the first time "new patients".
4. Patients who are willing to complete with the study requirements.
5. Patients who deny the blood sample will be included for the symptoms and risk factors analysis.
6. Patients who give written informed consent.

Exclusion Criteria:

1. Patients who will only be injected with BoNT once in our clinic at BCM.
2. Patients who deny participating in the clinical survey.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. The investigators plan to study 300 consecutive patients treated with BoNT at the Parkinson Disease center and Movement Disorders Clinic (PDCMDC) of Baylor College of Medicine.
  2. The investigators will invite patients to participate in the study during an eight-month period that includes two cycles of BoNT injections. All patients within this period will be invited to take part in the clinical study. This will include patients who have never been injected in our clinic and are considered as "new" patients; and patients who are followed on a regular basis in our clinic and are considered as "established" patients.
Sampling Method: Probability Sample
Enrollment: 247 (Actual)
Dates: Start 2011-04; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
The frequency of FLS will be estimated by number of patients and number of Botox treatments | Eight months or 2 treatment cycles
  The frequency of FLS will be estimated by number of patients and number of Botox treatments

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Jankovic, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Dept. of Neurology, Houston, Texas, United States